CLINICAL TRIAL: NCT03341728
Title: The Sensorimotor Locus of Balance Control in Elderly Gait
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 15-2267; R56AG054797-01A1 (NIH)
Record Dates: First submitted 2017-10-31; First posted 2017-11-14 (Actual); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-02

CONDITIONS: Ambulation Difficulty; Gait, Unsteady; Fall; Position Sense Disorders
MeSH Terms: conditions — Mobility Limitation; Gait Disorders, Neurologic; Somatosensory Disorders

STUDY DESIGN:
Intervention Model Description: In two 20 min sessions, on different days in a randomized cross-over design, older adults will walk with ("treatment" session) and without ("control" session) prolonged exposure to optical flow perturbations.
Masking Description: No Masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention, then Control (Experimental): Older adults will walk during exposure to optical flow perturbations
  Interventions: Behavioral: Optical flow perturbations; Behavioral: Normal walking
- Control, then Intervention (Experimental): Older adults will walk normally (without optical flow perturbations)
  Interventions: Behavioral: Optical flow perturbations; Behavioral: Normal walking

INTERVENTIONS:
Behavioral: Optical flow perturbations — Continuous mediolateral (i.e., side-to-side) 20-minute perturbations of optical flow that elicit the visual perception of lateral imbalance via virtual reality during treadmill walking.
Behavioral: Normal walking — Usual treadmill walking without optical flow perturbations

SUMMARY:
The aging population is at an exceptionally high risk of debilitating falls, contributing significantly to reduced independence and quality of life. It remains extremely challenging to screen for falls risk, and programs designed to mitigate falls risk have only modestly influenced the sizeable portion of the aging population experiencing one or more falls annually. Balance control in standing and walking depends on integrating reliable sensory feedback and on planning and executing appropriate motor responses. Walking balance control is especially dynamic, requiring active and coordinated adjustments in posture (i.e., trunk stabilization) and foot placement from step to step. Accordingly, using a custom, immersive virtual environment, the investigators have shown that sensory (i.e., optical flow) perturbations, especially when applied during walking, elicit strong and persistent motor responses to preserve balance. Exciting pilot data suggest that these motor responses are remarkably more prevalent in old age, presumably governed by an increased reliance on vision for balance control. Additional pilot data suggest that prolonged exposure to these perturbations may effectively condition successful balance control strategies. Founded on these recent discoveries, and leveraging the increase reliance on vision for balance control in old age, the investigators stand at the forefront of a potentially transformative new approach for more effectively identifying and mitigating age-related falls risk. The investigator's overarching hypothesis is that optical flow perturbations, particularly when applied during walking, can effectively identify balance deficits due to aging and falls history and can subsequently condition the neuromechanics of successful balance control via training.

DETAILED DESCRIPTION:
Specific Aim 1. Investigate sensory, motor, and cognitive-motor mechanisms governing susceptibility to optical flow perturbations. Aging increases the reliance on vision for balance control. However, central and peripheral mechanisms underlying aging and falls history effects on the susceptibility to optical flow perturbations are unclear. Hypothesis 1: Entrainment to optical flow perturbations will correlate most strongly with visual dependence and decreased somatosensory function, alluding to an age-associated process of multi-sensory reweighting. Methods: Multivariate models will quantify the extent to which strategically-selected sensory (i.e., visual dependence via rod/frame test, somatosensory function), motor (i.e., rate of torque development, timed sit-to-stand) and cognitive-motor (i.e., interference) mechanisms underlie inter-individual differences in susceptibility to perturbations.

Specific Aim 2. Estimate the efficacy of prolonged optical flow perturbations to condition the neuromechanics of walking balance control in older adult fallers. Pilot data from young adults suggests that prolonged exposure to optical flow perturbations may condition reactive strategies used to successfully control walking balance. The investigator's premise is that dynamic perturbation training can improve resilience to unexpected balance disturbances. Here, the investigators conduct a preliminary test of the effects of training with optical flow perturbations on walking balance in older adult fallers. Hypothesis 2: (a) Older adults with a history of falls will adapt to prolonged exposure to perturbations, conditioning their step to step adjustments in walking balance control, and (b) improving their response to unexpected balance challenges following training. Methods: In two 20 min sessions, on different days in a randomized cross-over design, older adults with a history of falls will walk with ("treatment" session) and without ("control" session) prolonged exposure to optical flow perturbations. The investigators will assess time-dependent changes in the neuromechanics of walking balance during training and after-effects via gait variability, dynamic stability, and performance on a series of real-world like targeting and obstacle avoidance tasks.

ELIGIBILITY:
Inclusion Criteria:

* Be able to walk without an assistive aid (i.e., walker, cane)
* Have the full capacity to provide informed consent

OLDER NON-FALLERS

* Age 65+ years
* No history of falls* in the prior 12 months

OLDER ADULTS WITH A HISTORY OF FALLS

* Age 65+ years
* History of one or more falls* in the prior 12 months

  * For the purposes of this study, falls counted towards the self-reported total will be defined as per the Kellogg International Work Group - a fall is "unintentionally coming to the ground or some lower level and other than as a consequence of sustaining a violent blow, loss of consciousness, sudden onset of paralysis as in stroke or an epileptic seizure"

Exclusion Criteria:

* Current lower extremity injury or fracture
* Taking medication that causes dizziness
* Have a leg prosthesis
* Prisoners
* Individuals clearly lacking the capacity to provide informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2018-07-25 (Actual); Study Completion 2018-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Franz, PhD, Principal Investigator — Unviersity of North Carolina at Chapel Hill
Locations (1):
- Applied Biomechanics Laboratory, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with other researchers.

REFERENCES:
- [Result] Franz JR, Francis CA, Allen MS, O'Connor SM, Thelen DG. Advanced age brings a greater reliance on visual feedback to maintain balance during walking. Hum Mov Sci. 2015 Apr;40:381-92. doi: 10.1016/j.humov.2015.01.012. Epub 2015 Feb 14. PMID 25687664
- [Result] Francis CA, Franz JR, O'Connor SM, Thelen DG. Gait variability in healthy old adults is more affected by a visual perturbation than by a cognitive or narrow step placement demand. Gait Posture. 2015 Sep;42(3):380-5. doi: 10.1016/j.gaitpost.2015.07.006. Epub 2015 Jul 17. PMID 26233581
- [Result] Thompson JD, Franz JR. Do kinematic metrics of walking balance adapt to perturbed optical flow? Hum Mov Sci. 2017 Aug;54:34-40. doi: 10.1016/j.humov.2017.03.004. Epub 2017 Apr 2. PMID 28371662
- [Result] Stokes HE, Thompson JD, Franz JR. The Neuromuscular Origins of Kinematic Variability during Perturbed Walking. Sci Rep. 2017 Apr 11;7(1):808. doi: 10.1038/s41598-017-00942-x. PMID 28400615
- [Derived] Richards JT, Selgrade BP, Qiao M, Plummer P, Wikstrom EA, Franz JR. Time-dependent tuning of balance control and aftereffects following optical flow perturbation training in older adults. J Neuroeng Rehabil. 2019 Jul 1;16(1):81. doi: 10.1186/s12984-019-0555-3. PMID 31262319
- See also: Applied Biomechanics Laboratory — http://abl.bme.unc.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention, Then Control: Older adults will first walk during exposure to optical flow perturbations
  Optical flow perturbations: Continuous mediolateral (i.e., side-to-side) 20-minute perturbations of optical flow that elicit the visual perception of lateral imbalance via virtual reality.
  Normal walking
- Control, Then Intervention: Older adults will first walk normally (without optical flow perturbations)
  Optical flow perturbations: Continuous mediolateral (i.e., side-to-side) 20-minute perturbations of optical flow that elicit the visual perception of lateral imbalance via virtual reality.
  Normal walking
Period: Session 1
Arm/Group | Intervention, Then Control | Control, Then Intervention
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0
Period: Washout (1 Week)
Arm/Group | Intervention, Then Control | Control, Then Intervention
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0
Period: Session 2
Arm/Group | Intervention, Then Control | Control, Then Intervention
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Older adults will walk during exposure to optical flow perturbations
  Optical flow perturbations: Continuous mediolateral (i.e., side-to-side) 20-minute perturbations of optical flow that elicit the visual perception of lateral imbalance via virtual reality.
  Normal walking
Arm/Group | All Participants
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14
History of Falls [Count of Participants; unit: Participants] — Self-reported history of at least 1 fall in the prior 12 months.
  Participants | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Postural Sway After 10 Min of Walking
Description: Magnitude of side-to-side postural sway
Time Frame: Baseline, 10 minutes
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Intervention: Older adults will walk during exposure to optical flow perturbations
  Optical flow perturbations: Continuous mediolateral (i.e., side-to-side) 20-minute perturbations of optical flow that elicit the visual perception of lateral imbalance via virtual reality.
- Normal Walking (Control): Older adults will first walk normally (without optical flow perturbations)
Arm/Group | Intervention | Normal Walking (Control)
Number analyzed (Participants) | 14 | 14
cm | -2.39 (1.10) | -0.01 (0.59)

2. Primary Outcome: Change in Kinematic Variability After 10 Min of Walking
Description: Magnitude of step-to-step corrections in step width measured in cm
Time Frame: Baseline, 10 minutes
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Intervention | Normal Walking (Control)
Number analyzed (Participants) | 14 | 14
cm | 0.55 (0.35) | 0.00 (0.01)

3. Primary Outcome: Change in Foot Placement Targeting Accuracy After 10 Min of Walking
Description: Accuracy of performing foot placement targeting task. i.e., distance between heel marker at initial contact and target line (measured using three-dimensional motion capture during walking).
Time Frame: Baseline, 10 minutes
Population: Data could not be collected because motion capture markers tracking the location of the targeting device were too often obstructed to be able to reliably estimate foot placement targeting accuracy.
Arm/Group | Intervention | Normal Walking (Control)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Cognitive-motor Interference Accuracy After 10 Min of Walking
Description: Accuracy performing an auditory stroop test (cognitive dual-task)
Time Frame: Baseline, 10 minutes
Population: Data could not be collected because noise from the treadmill motor interfered with the collection of auditory stroop test responses.
Arm/Group | Intervention | Normal Walking (Control)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Cognitive-motor Interference Response Time After 10 Min of Walking
Description: Response time in performing an auditory stroop test (cognitive dual-task)
Time Frame: Baseline, 10 minutes
Population: as for outcome 4
Arm/Group | Intervention | Normal Walking (Control)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Margin of Stability Variability After 10 Min of Walking
Description: Change in step-to-step fluctuations in margin of stability (the distance between the lateral boundary of the foot and the body's center of mass, measured in cm)
Time Frame: Baseline, 10 minutes
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Intervention | Normal Walking (Control)
Number analyzed (Participants) | 14 | 14
cm | -1.02 (0.99) | 0.16 (0.26)

ADVERSE EVENTS:
Time Frame: From the time of enrollment through the completion of the second 3-hour session approximately 1 week later
Arm/Group | Intervention | Normal Walking (Control)
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-01): https://cdn.clinicaltrials.gov/large-docs/28/NCT03341728/Prot_SAP_000.pdf